CLINICAL TRIAL: NCT06453356
Title: A PHASE 1 SINGLE INTRANASAL DOSE, OPEN-LABEL PHARMACOKINETIC STUDY OF ZAVEGEPANT IN HEALTHY LACTATING WOMEN
Brief Title: A Study to Learn How the Study Medicine Called Zavegepant is Taken Up Into Blood and Breast Milk of Healthy Breast-Feeding Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C5301032
Record Dates: First submitted 2024-05-28; First posted 2024-06-11 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zavegepant 10mg (Experimental): Intranasal (IN) 10mg spray on Day 1
  Interventions: Drug: Zavegepant 10mg

INTERVENTIONS:
Drug: Zavegepant 10mg — intransal spray 10mg
  Other Names: Zavzpret; PF-07930207

SUMMARY:
The purpose of the study is to look at the amount of zavegepant that is present in breast milk after single dose of zavegepant is sprayed through the nose in healthy breast-feeding women. This would allow to see if there are any possible risk to infants from medicines during breast-feeding.

The study is seeking for about 12 healthy breast-feeding females who are:

* 18 to 55 years of age.
* actively breast-feeding or producing breast milk.
* at least 2 weeks post-partum and not pregnant at present. Participants will not be allowed to breast-feed their infant from the evening of the day before to the first dose till 48 hours (2 days) after the dose.

Eligible participants will check into the clinical research unit (CRU) on Day -1. Participants will receive the zavegepant dose sprayed into the nose at the CRU on Day 1. The participants will stay at the CRU until the morning of Day 2. There will be collections of breast milk and plasma over 24 hours. Participants will be sent from the CRU on Day 2 and may begin to breastfeed their infant 48 hours (2 days) after the dose. A safety follow-up call will be done at about 28 to 35 days from the day the first dose of study medicine was given.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following key inclusion criteria to be eligible for enrollment into the study:

Age and Sex:

1. Healthy lactating females who are actively breast-feeding or expressing breast milk, who are at least 2 weeks post-partum and not currently pregnant (must have a negative pregnancy test), and must be 18 to 55 years of age, inclusive, at the time of signing the Informed Consent Document (ICD).

   • Participants must be able to express at least 14 mL of breast milk over a 2-hour interval prior to the dose on Day 1.

   Other Inclusion Criteria:
2. Body mass index (BMI) 16.0-34.9 kg/m2 and body weight ≥45.0 kg (99 lb).
3. Female participants with history of acute migraine are allowed.
4. Participants must be willing to temporarily discontinue breastfeeding their infants for a total of 2.5 days (approximately 60 hours), ie, from the evening of the day before Day 1 through to 48 hours after the dose (approximately 8 AM the morning of Day 3). Participants must be willing to regularly pump breasts throughout the study and express breast milk according to a schedule designed to maintain lactation throughout the study period.
5. Participants must agree that breast milk expressed following zavegepant administration through 48 hours after the dose should be discarded and will not be fed to any infant.

   -

Exclusion Criteria:

Participants with any of the following characteristics/conditions will be excluded:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological (with exception of acute migraine), or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Clinically significant history of nasal conditions that may affect the administration or absorption of the nasal product (eg, severe septum deviation or nasal deformity, inflammation, perforation, mucosal erosion or ulceration, localized infection, congestion, polyposis, rhinorrhea, nasal surgery within the previous 6 months, or nasal trauma).
3. Significant history of seizure disorder other than a single childhood febrile seizure (eg, epilepsy).
4. History of gallstone or cholecystectomy.
5. Any other medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to coronavirus disease 2019 (COVID-19) pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
6. Use of organic anion transporting polypeptide 1B3 (OATP1B3) inhibitors within 14 days or 5 half-lives, whichever is longer, before first dosing.
7. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to investigational product (IP) dosing, administration of a biological product in the context of a clinical research study within 90 days prior to IP dosing, or concomitant participation in an investigational study involving no drug or device administration.
8. Any clinically significant abnormal laboratory test results or positive test found during medical screening. A single repeat for positive drug screen may be allowed at the discretion of the principal investigator (PI).
9. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination or nasal inspection beyond what is consistent with the target population.
10. Participants with ANY of the following abnormalities in clinical laboratory tests at screening:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level > 1.5 × upper limit of normal (ULN);
    * Total bilirubin level >1.5 × ULN;
    * Estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73m².
11. Individuals who smoke more than 5 cigarettes or equivalent daily.
12. Presence of piercings or any physical findings in the nose that, in the opinion of the PI, would likely interfere with the successful completion of the dosing procedure.
13. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
14. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
15. Any reason that, in the opinion of the PI, would prevent the participant from participating in the study.

    -

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Area Under the Breast Milk Concentration-time Profile from time 0 extrapolated to infinite time (AUCinf), if data permit | 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 16, 16 to 24 hours
  AUCinf = Area under the breast milk concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Area Under the Breast Milk Concentration-time Profile From Time Zero to the Time of Last Quantifiable Concentration (AUClast) | 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 16, 16 to 24 hours
  Area under the breast milk concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Breast Milk Concentration-time Profile From Time Zero to the Time of 24 hr post dose (AUC24) | 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 16, 16 to 24 hours
  AUC24= Area under the breast milk concentration versus time curve from time zero (pre-dose) to time 24 hours
Maximum observed breast milk concentration (Cmax) | 0 to 24 hours post dose
Time for Cmax in Breast Milk (Tmax) | 0 to 24 hours post dose
Terminal half-life for breast milk (t 1/2), if data permit | 0 to 24 hours post dose

SECONDARY OUTCOMES:
Area under the concentration-time profile from time 0 extrapolated to infinite time (AUCinf), if data permit | 0 to 24 hours post dose
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Area under the concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast) | 0 to 24 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area under the concentration-time profile from time 0 to 24 hours post dose (AUC24) | 0 to 24 hours post dose
  AUC24= Area under the plasma concentration versus time curve from time zero (pre-dose) to time 24 hours
Maximum observed plasma concentration (Cmax) | 0 to 24 hours post dose
Time for plasma Cmax (Tmax) | 0 to 24 hours post dose
Plasma Terminal half-life (t 1/2), if data permit | 0 to 24 hours post dose
Average plasma concentration (Cav) over 24 hr | 0 to 24 hours post dose
Breast milk to plasma ratio for AUCinf (MPAUCinf), if data permit | 0 to 24 hours post dose
Breast milk to plasma ratio (MPAUC24) for AUC24, if data permit | 0 to 24 hours post dose
Breast milk to plasma ratio for Cmax (MPCmax) | 0 to 24 hours post dose
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From Day 1 up to at least 28 days after last dose of study drug
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | 0 to 24 hours post dose
Number of Participants With Clinically Significant Change from Baseline in Electrocardiogram (ECG) Parameters | 0 to 24 hours post dose
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | 0 to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO, Springfield, Missouri
  - Bio-Kinetic Clinicals Applications LLC DBA QPS-MO Patient Screening and Recruitment Center Center), Springfield, Missouri

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5301032